CLINICAL TRIAL: NCT06484088
Title: Characterizing the Brain Circuitry and Neural Activity Mediating Frustration
Brief Title: Study Brain Mechanisms of Frustration With Magnetoencephalography in Healthy Volunteers
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10002073; 002073-M
Record Dates: First submitted 2024-06-29; First posted 2024-07-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01-27

CONDITIONS: Irritability
Keywords: Healthy volunteers, Frustration, Magnetoencephalography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frustration task (Experimental): The experimental manipulation for this study is the frustration task. The frustration task is designed to elicit the emotional state of frustrative non-reward (FNR). During the task, participants are asked to use button press (left or right) to alternately press one of the two doors displayed on the monitor. The task has two non-frustration blocks (Block 1 and 2) and one frustration block (Block 3). During the non-frustration blocks, participants earn money for correct press on a fixed schedule. During the frustrative block, participants will not always receive reward for correct press.
  Interventions: Other: Frustration task

INTERVENTIONS:
Other: Frustration task — The experimental manipulation for this study is the frustration task. The frustration task is designed to elicit the emotional state of frustrative non-reward (FNR). During the task, participants are asked to use button press (left or right) to alternately press one of the two doors displayed on the monitor. The task has two non-frustration blocks (Block 1 and 2) and one frustration block (Block 3). During the non-frustration blocks, participants earn money for correct press on a fixed schedule. During the frustrative block, participants will not always receive reward for correct press.

SUMMARY:
Background:

Irritability can be defined as an unusually strong response to frustration; these responses may include severe temper outbursts and a constant grumpy mood. Irritability is a common symptom of many mental health disorders. Little is known about how the brain responds to frustration, and few treatments are available for this problem. Researchers want to know more about how the brain responds to frustration.

Objective:

To learn how the brain responds to frustration.

Eligibility:

Healthy adults aged 18 to 55 years. They must have been screened through studies 01-M-0254 or 17-M-0181.

Design:

Participants will have up to 3 study visits in 2 months. Each visit will last up to 4 hours.

Visit 1: Participants will be screened. They will have a physical exam. They will complete questionnaires about how often and how easily they get angry or grumpy. They will be trained to use a device that measures hand grip.

Visit 2: Participants will have a magnetic resonance imaging (MRI) scan. They will lie on a table that slides into a tube. Padding will hold their head still.

Visit 3: Participants will undergo magnetoencephalography (MEG). A cone with detectors will be lowered over their head while they are seated. The MEG will measure the magnetic fields in the participant s brain both while they are resting and while they are doing the frustration task. For the task, they will hold a grip device in each hand. They will use the devices to pick 1 of 2 doors on a computer screen. The task has 3 parts. The participant s face will be filmed during this task.

DETAILED DESCRIPTION:
STUDY DESCRIPTION:

Participants in this study will be healthy adults. This protocol uses a frustration induction task, magnetoencephalography (MEG), and brain magnetic resonance imaging (MRI), coupled with physical and self-report assessment of frustration, to study brain mechanisms underlying frustration in adults. This study is part of a cross-species project; hence, hypotheses are based on neural mechanisms of frustration identified in mice.

OBJECTIVES:

To use a frustration induction task, MEG, and brain MRI, coupled with physical and self-report assessment of frustration, to measure how frustration alters synchronized neural activities and physical activities. Specifically, we will identify brain circuits and neural oscillations that potentially underly the emotional and behavioral consequences of frustration and characteristic changes in grip force, pupil/cornea size, and facial expressions that can be used as objective measurements of frustration.

ENDPOINTS:

1. The power of neural oscillations in the cortical-basal gangliathalamic circuit, which we hypothesize will be altered by frustration comparing pre and post-frustration resting states, and increased more by unexpected reward omission than reward attainment;
2. Coherence of neural oscillations in the above-mentioned circuit, which we hypothesize will be increased in the beta band by unexpected reward omission but not by expected reward omission, and that this decrease will accumulate with the number of frustration episodes; (3) Frustration rating by self-report, facial expression, pupil/cornea size, and the duration and strength of gripping, which we hypothesize will be higher after unexpected reward omission than after expected reward omission

ELIGIBILITY:
-INCLUSION CRITERIA:

This study will include adult healthy volunteers.

* Age: 18-55
* Consent: can give consent
* Speak and read English

  --The instruments have not been validated in other languages.
* At the NIH site, previously screened through other NIH protocols such as protocol 01-M-0254, 17-M-0181, and 93-M-0170 and determined eligible as healthy volunteers.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

-Any serious medical condition

* History, physical exam, or laboratory testing including drug abuse screen.

  -Prescription and over-the-counter medications and dietary supplements with psychoactive properties (e.g., St. John's Wort, Melatonin, Valerian)

  -Any condition that interferes with MRI or MEG**
* History

  -Any current psychiatric diagnosis
* SCID-V, clinical assessment, or history.

  -Pregnancy
* Pregnancy testing will be done before all MRIs.

  -People who work on night shifts
* History

  -Drug use
* Subjects with drug use or positive drug screen more than two years ago are eligible for participation.

  -Need to wear eye glasses to work with computers*
* History

  -Need to wear contact lenses to work with computers**,***
* History

  -Dental retainer**
* Subjects wearing removable dental retainers are eligible for participation

  * Eye glasses create artifacts in MEG and their rigid shape does not fit well in the MEG scanner. The MEG core has plastic optometry lenses that can be placed in paper frames. However, the paper frames need to be secured with tape which makes wearing them very uncomfortable, potentially promoting negative emotion and reducing the reliability of facial expression analysis.

    * Only applies to the NIH site.

      * Contact lenses create artifacts that interfere with eye-tracking.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
(1) The power of neural oscillations in the cortical-basal ganglia-thalamic circuit; (2) Coherence of neural oscillations in this circuit; (3) Frustration rating by self-report, facial expression, and the duration and strength of gripping. | The measurements will be taken during the MEG/frustration task session.
  MEG recording is acquired during the frustration task. 3-6 minutes of resting-state recording is acquired before, between, and after each block of the frustration task. Feelings of frustration and unhappiness were assessed after each run using 9-point Likert scales. Frustration assessment takes place before and after the task and between each block within the task. The strength and duration of gripping the press device during the task is recorded for all trials.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Li, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Texas A&M University, College Station, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies results in a publication will be made available upon requested by other researchers. If participants are co-enrolled in another NIH protocol, then data collected in either study may be shared with and used for research in either study.
Supporting Information: SAP
Time Frame: IPD that under results in a publication may be requested by other researchers when the publication is online or in print or by the end of the project/protocol, whichever comes first.
Access Criteria: IPD that under results in a publication will be made public through NIH-supported scientific data repositories. Access criteria are defined by the repositories and not limited by analysis type.

REFERENCES:
- [Background] Beauchaine TP, Tackett JL. Irritability as a Transdiagnostic Vulnerability Trait:Current Issues and Future Directions. Behav Ther. 2020 Mar;51(2):350-364. doi: 10.1016/j.beth.2019.10.009. Epub 2019 Nov 27. PMID 32138943
- [Background] Brotman MA, Kircanski K, Leibenluft E. Irritability in Children and Adolescents. Annu Rev Clin Psychol. 2017 May 8;13:317-341. doi: 10.1146/annurev-clinpsy-032816-044941. PMID 28482689
- [Background] Eshel N, Leibenluft E. New Frontiers in Irritability Research-From Cradle to Grave and Bench to Bedside. JAMA Psychiatry. 2020 Mar 1;77(3):227-228. doi: 10.1001/jamapsychiatry.2019.3686. No abstract available. PMID 31799997
- [Background] Linke JO, Haller SP, Xu EP, Nguyen LT, Chue AE, Botz-Zapp C, Revzina O, Perlstein S, Ross AJ, Tseng WL, Shaw P, Brotman MA, Pine DS, Gotts SJ, Leibenluft E, Kircanski K. Persistent Frustration-Induced Reconfigurations of Brain Networks Predict Individual Differences in Irritability. J Am Acad Child Adolesc Psychiatry. 2023 Jun;62(6):684-695. doi: 10.1016/j.jaac.2022.11.009. Epub 2022 Dec 21. PMID 36563874
- [Background] Tseng WL, Deveney CM, Stoddard J, Kircanski K, Frackman AE, Yi JY, Hsu D, Moroney E, Machlin L, Donahue L, Roule A, Perhamus G, Reynolds RC, Roberson-Nay R, Hettema JM, Towbin KE, Stringaris A, Pine DS, Brotman MA, Leibenluft E. Brain Mechanisms of Attention Orienting Following Frustration: Associations With Irritability and Age in Youths. Am J Psychiatry. 2019 Jan 1;176(1):67-76. doi: 10.1176/appi.ajp.2018.18040491. Epub 2018 Oct 19. PMID 30336704
- [Background] AMSEL A. The role of frustrative nonreward in noncontinuous reward situations. Psychol Bull. 1958 Mar;55(2):102-19. doi: 10.1037/h0043125. No abstract available. PMID 13527595
- [Background] Naik AA, Ma X, Munyeshyaka M, Leibenluft E, Li Z. A New Behavioral Paradigm for Frustrative Non-reward Reveals a Global Change in Brain Networks by Frustration. bioRxiv [Preprint]. 2023 Jun 6:2023.02.28.530477. doi: 10.1101/2023.02.28.530477. PMID 36909498
- [Background] Naik AA, Ma X, Munyeshyaka M, Leibenluft E, Li Z. A New Behavioral Paradigm for Frustrative Nonreward in Juvenile Mice. Biol Psychiatry Glob Open Sci. 2023 Nov 17;4(1):31-38. doi: 10.1016/j.bpsgos.2023.09.007. eCollection 2024 Jan. PMID 38045768
- [Background] Vrba J, Robinson SE. Signal processing in magnetoencephalography. Methods. 2001 Oct;25(2):249-71. doi: 10.1006/meth.2001.1238. PMID 11812209
- [Background] Pizzo F, Roehri N, Medina Villalon S, Trebuchon A, Chen S, Lagarde S, Carron R, Gavaret M, Giusiano B, McGonigal A, Bartolomei F, Badier JM, Benar CG. Deep brain activities can be detected with magnetoencephalography. Nat Commun. 2019 Feb 27;10(1):971. doi: 10.1038/s41467-019-08665-5. PMID 30814498
- [Background] Salvadore G, Cornwell BR, Sambataro F, Latov D, Colon-Rosario V, Carver F, Holroyd T, DiazGranados N, Machado-Vieira R, Grillon C, Drevets WC, Zarate CA Jr. Anterior cingulate desynchronization and functional connectivity with the amygdala during a working memory task predict rapid antidepressant response to ketamine. Neuropsychopharmacology. 2010 Jun;35(7):1415-22. doi: 10.1038/npp.2010.24. Epub 2010 Mar 10. PMID 20393460
- [Background] Cornwell BR, Carver FW, Coppola R, Johnson L, Alvarez R, Grillon C. Evoked amygdala responses to negative faces revealed by adaptive MEG beamformers. Brain Res. 2008 Dec 9;1244:103-12. doi: 10.1016/j.brainres.2008.09.068. Epub 2008 Oct 7. PMID 18930036
- [Background] Carlson GA, Singh MK. Emotion Dysregulation and Outbursts in Children and Adolescents: Part I. Child Adolesc Psychiatr Clin N Am. 2021 Apr;30(2):xiii-xvi. doi: 10.1016/j.chc.2020.10.014. Epub 2021 Feb 15. No abstract available. PMID 33743952
- [Background] Singh MK, Carlson GA. Emotion Dysregulation in Children and Adolescents: Part II. Child Adolesc Psychiatr Clin N Am. 2021 Jul;30(3):xiii-xiv. doi: 10.1016/j.chc.2021.05.002. No abstract available. PMID 34053694
- [Background] Tseng WL, Naim R, Chue A, Shaughnessy S, Meigs J, Pine DS, Leibenluft E, Kircanski K, Brotman MA. Network analysis of ecological momentary assessment identifies frustration as a central node in irritability. J Child Psychol Psychiatry. 2023 Aug;64(8):1212-1221. doi: 10.1111/jcpp.13794. Epub 2023 Mar 28. PMID 36977629
- [Background] Abler B, Walter H, Erk S. Neural correlates of frustration. Neuroreport. 2005 May 12;16(7):669-72. doi: 10.1097/00001756-200505120-00003. PMID 15858403
- [Background] Bierzynska M, Bielecki M, Marchewka A, Debowska W, Duszyk A, Zajkowski W, Falkiewicz M, Nowicka A, Strelau J, Kossut M. Effect of Frustration on Brain Activation Pattern in Subjects with Different Temperament. Front Psychol. 2016 Jan 11;6:1989. doi: 10.3389/fpsyg.2015.01989. eCollection 2015. PMID 26793136
- [Background] Deveney CM, Connolly ME, Haring CT, Bones BL, Reynolds RC, Kim P, Pine DS, Leibenluft E. Neural mechanisms of frustration in chronically irritable children. Am J Psychiatry. 2013 Oct;170(10):1186-94. doi: 10.1176/appi.ajp.2013.12070917. PMID 23732841
- [Background] Grabell AS, Li Y, Barker JW, Wakschlag LS, Huppert TJ, Perlman SB. Evidence of Non-Linear Associations between Frustration-Related Prefrontal Cortex Activation and the Normal:Abnormal Spectrum of Irritability in Young Children. J Abnorm Child Psychol. 2018 Jan;46(1):137-147. doi: 10.1007/s10802-017-0286-5. PMID 28315125
- [Background] Pawliczek CM, Derntl B, Kellermann T, Gur RC, Schneider F, Habel U. Anger under control: neural correlates of frustration as a function of trait aggression. PLoS One. 2013 Oct 18;8(10):e78503. doi: 10.1371/journal.pone.0078503. eCollection 2013. PMID 24205247
- [Background] Perlman SB, Jones BM, Wakschlag LS, Axelson D, Birmaher B, Phillips ML. Neural substrates of child irritability in typically developing and psychiatric populations. Dev Cogn Neurosci. 2015 Aug;14:71-80. doi: 10.1016/j.dcn.2015.07.003. Epub 2015 Jul 20. PMID 26218424
- [Background] Rich BA, Holroyd T, Carver FW, Onelio LM, Mendoza JK, Cornwell BR, Fox NA, Pine DS, Coppola R, Leibenluft E. A preliminary study of the neural mechanisms of frustration in pediatric bipolar disorder using magnetoencephalography. Depress Anxiety. 2010 Mar;27(3):276-86. doi: 10.1002/da.20649. PMID 20037920
- [Background] Yu R, Mobbs D, Seymour B, Rowe JB, Calder AJ. The neural signature of escalating frustration in humans. Cortex. 2014 May;54:165-78. doi: 10.1016/j.cortex.2014.02.013. Epub 2014 Mar 11. PMID 24699035
- [Background] AMSEL A, HANCOCK W. Motivational properties of frustration. III. Relation of frustration effect to antedating goal factors. J Exp Psychol. 1957 Feb;53(2):126-31. doi: 10.1037/h0042075. No abstract available. PMID 13406193
- [Background] Brotman MA, Kircanski K, Stringaris A, Pine DS, Leibenluft E. Irritability in Youths: A Translational Model. Am J Psychiatry. 2017 Jun 1;174(6):520-532. doi: 10.1176/appi.ajp.2016.16070839. Epub 2017 Jan 20. PMID 28103715
- [Background] Morgan JI, Cohen DR, Hempstead JL, Curran T. Mapping patterns of c-fos expression in the central nervous system after seizure. Science. 1987 Jul 10;237(4811):192-7. doi: 10.1126/science.3037702.
- [Background] Sheng M, Greenberg ME. The regulation and function of c-fos and other immediate early genes in the nervous system. Neuron. 1990 Apr;4(4):477-85. doi: 10.1016/0896-6273(90)90106-p. No abstract available. PMID 1969743
- [Background] Post RJ, Bulkin DA, Ebitz RB, Lee V, Han K, Warden MR. Tonic activity in lateral habenula neurons acts as a neutral valence brake on reward-seeking behavior. Curr Biol. 2022 Oct 24;32(20):4325-4336.e5. doi: 10.1016/j.cub.2022.08.016. Epub 2022 Aug 31. PMID 36049479
- [Background] Starkweather CK, Uchida N. Dopamine signals as temporal difference errors: recent advances. Curr Opin Neurobiol. 2021 Apr;67:95-105. doi: 10.1016/j.conb.2020.08.014. Epub 2020 Nov 10. PMID 33186815
- [Background] Haber SN, Knutson B. The reward circuit: linking primate anatomy and human imaging. Neuropsychopharmacology. 2010 Jan;35(1):4-26. doi: 10.1038/npp.2009.129. PMID 19812543
- [Background] Dugre JR, Potvin S. Neural bases of frustration-aggression theory: A multi-domain meta-analysis of functional neuroimaging studies. J Affect Disord. 2023 Jun 15;331:64-76. doi: 10.1016/j.jad.2023.03.005. Epub 2023 Mar 15. PMID 36924847
- [Background] Scheinost D, Dadashkarimi J, Finn ES, Wambach CG, MacGillivray C, Roule AL, Niendam TA, Pine DS, Brotman MA, Leibenluft E, Tseng WL. Functional connectivity during frustration: a preliminary study of predictive modeling of irritability in youth. Neuropsychopharmacology. 2021 Jun;46(7):1300-1306. doi: 10.1038/s41386-020-00954-8. Epub 2021 Jan 21. PMID 33479511
- [Background] Leibenluft E, Allen LE, Althoff RR, Brotman MA, Burke JD, Carlson GA, Dickstein DP, Dougherty LR, Evans SC, Kircanski K, Klein DN, Malone EP, Mazefsky CA, Nigg J, Perlman SB, Pine DS, Roy AK, Salum GA, Shakeshaft A, Silver J, Stoddard J, Thapar A, Tseng WL, Vidal-Ribas P, Wakschlag LS, Stringaris A. Irritability in Youths: A Critical Integrative Review. Am J Psychiatry. 2024 Apr 1;181(4):275-290. doi: 10.1176/appi.ajp.20230256. Epub 2024 Feb 29. PMID 38419494
- [Background] Haller SP, Kircanski K, Stringaris A, Clayton M, Bui H, Agorsor C, Cardenas SI, Towbin KE, Pine DS, Leibenluft E, Brotman MA. The Clinician Affective Reactivity Index: Validity and Reliability of a Clinician-Rated Assessment of Irritability. Behav Ther. 2020 Mar;51(2):283-293. doi: 10.1016/j.beth.2019.10.005. Epub 2019 Nov 27. PMID 32138938
- [Background] Stringaris A, Goodman R, Ferdinando S, Razdan V, Muhrer E, Leibenluft E, Brotman MA. The Affective Reactivity Index: a concise irritability scale for clinical and research settings. J Child Psychol Psychiatry. 2012 Nov;53(11):1109-17. doi: 10.1111/j.1469-7610.2012.02561.x. Epub 2012 May 10. PMID 22574736
- [Background] Holtzman S, O'Connor BP, Barata PC, Stewart DE. The Brief Irritability Test (BITe): a measure of irritability for use among men and women. Assessment. 2015 Feb;22(1):101-15. doi: 10.1177/1073191114533814. Epub 2014 May 15. PMID 24830513
- [Background] Staddon JE, Cerutti DT. Operant conditioning. Annu Rev Psychol. 2003;54:115-44. doi: 10.1146/annurev.psych.54.101601.145124. Epub 2002 Jun 10. PMID 12415075
- [Background] Vasquez TES, Shah P, Re JD, Laezza F, Green TA. Individual Differences in Frustrative Nonreward Behavior for Sucrose in Rats Predict Motivation for Fentanyl under Progressive Ratio. eNeuro. 2021 Oct 27;8(5):ENEURO.0136-21.2021. doi: 10.1523/ENEURO.0136-21.2021. Print 2021 Sep-Oct. PMID 34607807
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002073-M.html